CLINICAL TRIAL: NCT03892278
Title: Effects of 16 Weeks of Different Water-based Training Programs on Neuromuscular, Cardiorespiratory, Functional Capacity, Quality of Life and Cognitive Function Variables in Elderly Woman: a Randomized Clinical Trial
Brief Title: Effects of Water-based Aerobic and Combined Training in Elderly Woman
Acronym: ACTIVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Stephanie Santana Pinto, Professor in physical education school, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTIVE
Record Dates: First submitted 2019-03-05; First posted 2019-03-27 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Elderly Women
Keywords: combined training; aerobic training; aquatic exercises; aging
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic training (Experimental): Participants who will be randomized for the intervention in the aerobic training group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle and participants will carry out three 3-minute series of each exercise. In the first mesocycle (weeks 1-2) the intensity will correspond to 80-85% of heart rate corresponding to the anaerobic threshold (HRat). In the second mesocycle (weeks 3-4) the intensity will correspond to 85-90% of HRat. In the third mesocycle, the intensity will correspond to 90-95% of HRat from weeks 5-7. In the fourth mesocycle, the intensity will correspond to 95-100% of HRat from weeks 8-10. In the fifth mesocycle (weeks 11-13) the intensity will correspond to the 100-105% of HRat for 2 minutes and <85% of HRat for 1 minute. The last mesocycle (weeks 14-16) the intensity will correspond to the 105-110% of HRat for 2 minutes and <85% of HRat for 1 minute.
  Interventions: Behavioral: Water-based aerobic training
- Aerobic and combined training (Experimental): Participants who will be randomized for the intervention in the aerobic and combined training group will perform 8 weeks of aerobic training and more 8 weeks of aerobic and resistance training in same session. In aerobic training the participants will perform three 3-min series of each exercise. The intensity will correspond to 80-85% of heart rate of anaerobic threshold (HRat) (weeks 1-2), 85-90% of HRat (weeks 3-4), 90-95% of HRat (weeks 5-7), 95-100% of HRat (weeks 8-10), 100-105% for 2 min and <85% of HRat for 1 min (weeks 11-13) and 105-110% for 2 min and <85% of HRat for 1 min (weeks 14-16). Resistance training will be divide into two blocks of exercises perform each repetition at maximal effort, speed and amplitude. Participants will perform 2 sets of 30 s for each block in the first mesocycle (weeks 9-10), 3 sets of 20 s in the second mesocycle (weeks 11-13) and 4 sets of 15 s in the third mesocycle (weeks 14-16).
  Interventions: Behavioral: Water-based aerobic and combined training
- Control group (Active Comparator): The control group will perform a weekly session composed of 30 minutes of therapeutic and playfull exercises in the aquatic environment, involving games, relaxation, massage and conversation.The participants will receive instructions to perform the movements as slowly as possible to avoid physical effort.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Water-based aerobic training — Participants who will be randomized for the intervention in the aerobic training group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle and participants will carry out three 3-minute series of each exercise. In the first mesocycle (weeks 1-2) the intensity will correspond to 80-85% of heart rate corresponding to the anaerobic threshold (HRat). In the second mesocycle (weeks 3-4) the intensity will correspond to 85-90% of HRat. In the third mesocycle, the intensity will correspond to 90-95% of HRat from weeks 5-7. In the fourth mesocycle, the intensity will correspond to 95-100% of HRat from weeks 8-10. In the fifth mesocycle (weeks 11-13) the intensity will correspond to the 100-105% of HRat for 2 minutes and <85% of HRat for 1 minute. The last mesocycle (weeks 14-16) the intensity will correspond to the 105-110% of HRat for 2 minutes and <85% of HRat for 1 minute.
  Arms: Aerobic training
Behavioral: Water-based aerobic and combined training — Participants who will be randomized for the intervention in the aerobic and combined training group will perform 8 weeks of aerobic training and more 8 weeks of aerobic and resistance training in same session. In aerobic training the participants will perform three 3-min series of each exercise. The intensity will correspond to 80-85% of heart rate of anaerobic threshold (HRat) (weeks 1-2), 85-90% of HRat (weeks 3-4), 90-95% of HRat (weeks 5-7), 95-100% of HRat (weeks 8-10), 100-105% for 2 min and <85% of HRat for 1 min (weeks 11-13) and 105-110% for 2 min and <85% of HRat for 1 min (weeks 14-16). Resistance training will be divide into two blocks of exercises perform each repetition at maximal effort, speed and amplitude. Participants will perform 2 sets of 30 s for each block in the first mesocycle (weeks 9-10), 3 sets of 20 s in the second mesocycle (weeks 11-13) and 4 sets of 15 s in the third mesocycle (weeks 14-16).
  Arms: Aerobic and combined training
Behavioral: Control group — The control group will perform a weekly session composed of 30 minutes of therapeutic and playfull exercises in the aquatic environment, involving games, relaxation, massage and conversation.The participants will receive instructions to perform the movements as slowly as possible to avoid physical effort.
  Arms: Control group

SUMMARY:
Purpose: Investigate neuromuscular, cardiorespiratory, functional capacity, quality of life and cognitive adaptations of eight weeks of water-based aerobic and combined training in elderly women previously trained for eight weeks of water-based aerobic training.

Materials and methods: Fifty-four elderly women volunteer will be randomly divided into two groups with ratio of 2:1 (week 0): water-based aerobic training (WBA) and control group (CG). After eight weeks of intervention the WBA group will be randomly divided into two groups with ratio of 1:1 (week 9): WBA and water-based combined training (WBC). The intervention will last 16 weeks with two weekly sessions for water-based training groups and one weekly session for CG. The WBA program will consist only of aerobic exercises while the WBC program will consist of aerobic and resistance exercises in the same session. The WBA training will be performed in the percentages of heart rate corresponding to the anaerobic threshold and the resistance training sets will be performed at maximal effort. Assessments of muscular endurance of knee extensors and elbow flexors, peak oxygen consumption and ventilatory thresholds, occurrence of low back pain and disability from the same, functional capacity (30-second chair stand, 8-foot up-and-go and chair sit-and-reach) and of functional test 8-foot up-and-go with counting task will be performed before (week 0) and after interventions (week 17). Moreover, assessments of maximal dynamic strength in knee extensors and elbow flexors, maximal neuromuscular activity and maximal voluntary isometric contraction of knee extensor muscles, muscle thickness and echo intensity of knee extensor muscles, heart rate, blood pressure, functional capacity (6-minute walk), quality of life and cognitive function will be performed before (week 0), between (week 9) and after interventions (week 17). The data will be analyzed using Generalized Estimating Equations (GEE) and Bonferroni post-hoc test (α=0,05).

DETAILED DESCRIPTION:
Aging process has its own characteristics, among which the direct association with reductions in muscle mass, muscle strength and cardiorespiratory fitness are highlighted. These reductions cause impairment in functional capacity, affecting the efficiency of elderly individuals to perform daily living tasks. However regular exercise practice can be efficient to mitigate factors associated with aging.

A modality that has been well suited for individuals over 60 years is the water-based exercises training, precisely due to the beneficial conditions of the aquatic environment, such as the lower impact on the lower limbs joints in comparison to the impact observed during exercises performed on land

The aim of the study is to investigate neuromuscular, cardiorespiratory, functional capacity, quality of life and cognitive adaptations of eight weeks of water-based aerobic and combined training in elderly women previously trained for eight weeks of water-based aerobic training.

Volunteer old women age range: 60-75 years old, will participate to this study, and will randomly divided into three groups: water-based aerobic training group (WBA), water-based aerobic and combined training group (WBAC) and control group (CG).

Fifty-four elderly women volunteer will be randomly divided into two groups with ratio of 2:1 (week 0): WBA and CG. After eight weeks of intervention the WBA group will be randomly divided into two groups with ratio of 1:1 (week 9): WBA and water-based combined training (WBC).

The intervention will last 16 weeks with two weekly sessions for water-based training groups and one weekly session for CG. The WBA program will consist only of aerobic exercises while the WBC program will consist of aerobic and resistance exercises in the same session.

Participants who will be randomized for WBA group will carry out exercises with no interval for exercise change. Intensity will be increased every mesocycle. In the first mesocycle (weeks 1-2), participants will carry out three 3-minute series of each exercise whose intensity corresponds 80-85% of heart rate corresponding to the anaerobic threshold (HRat). In the second mesocycle (weeks 3-4), participants will perform three 3-minute series of each exercise corresponding to 85-90% of HRat. In the third mesocycle, participants will perform three 3-minute series of each exercise at intensity corresponding to 90-95% of HRat from weeks 5-7. In the fourth mesocycle, participants will perform three 3-minute series of each exercise at intensity corresponding to 95-100% of HRat from weeks 8-10. In the fifth mesocycle (weeks 11-13) comprises three 3-minute series of each exercise whose intensity corresponds to the 100-105% of HRat for 2 minutes and <85% of HRat for 1 minute. The last mesocycle (weeks 14-16) comprises three 3-minute series of each exercise whose intensity corresponds to the 105-110% of HRat for 2 minutes and <85% of HRat for 1 minute.

Resistance training will be divide into two blocks of exercises, and each block will be compose of one exercise for the upper and one for the lower limbs. Block 1 will consist of shoulder flexion and extension (bilateral) and hip flexion and extension (unilateral) exercises. Block 2 will consist of elbow flexion and extension (bilateral) and knee flexion and extension, starting from 90° of hip flexion (unilateral), exercises. In the first mesocycle (weeks 9-10) participants will perform 2 sets of 30 s for each block with the following sequence: 30 s of exercise for the lower limb (right leg), 5 s for switching, 30 s of exercise for the lower limb (left leg), 5 s for switching and 30 s of exercise for the upper limbs. The blocks sequences and intervals will be as follows: block 1 (4 min 20s), interval between blocks (1 min) and block 2 (4 min 20 s). In the second mesocycle (weeks 11-13) participants will perform 3 sets of 20 s for each block.The blocks sequences and intervals will be as follows: 3 times block 1 (6 min 10 s), interval between blocks (1 min) and block 2 (6 min 10 s). In the third mesocycle (weeks 14-16) the participants will perform 4 sets of 15 s for each block. The blocks sequences and intervals will be as follows: 4 times block 1 (8 min 10 s), interval between blocks (1 min) and 4 times block 2 (8 min 10 s).

Assessments of muscular endurance of knee extensors and elbow flexors, peak oxygen consumption and ventilatory thresholds, occurrence of low back pain and disability from the same, functional capacity (30-second chair stand, 8-foot up-and-go and chair sit-and-reach) and of functional test 8-foot up-and-go with counting task will be performed before (week 0) and after interventions (week 17). Moreover, assessments of maximal dynamic strength in knee extensors and elbow flexors, maximal neuromuscular activity and maximal voluntary isometric contraction of knee extensor muscles, muscle thickness and echo intensity of knee extensor muscles, heart rate, blood pressure, functional capacity (6-minute walk), quality of life and cognitive function will be performed before (week 0), between (week 9) and after interventions (week 17).

The data will be analyzed using Generalized Estimating Equations (GEE) and Bonferroni post-hoc test (α=0,05).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer elderly women, aged between 60-75 years old who were not participating on any regular training program in the last four months

Exclusion Criteria:

* Cardiovascular disease (except hypertension controlled by medication);
* Physical impairments for exercise diagnosed through anamnesis;

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Maximal dynamic strength change after eight and sixteen weeks (Kg) | Baseline, 8 week and 16 week
  Maximal dynamic strenght will be evaluate sing the one-repetition maximum test (1RM) on the bilateral knee extensors and free-weight barbell bilateral elbow flexors. The 1RM value will be consider as the maximal load that could be exerted at the concentric phase for a given exercise. Subjects will be familiar with al procedures in a session one week prior to the test day. Performance time for each contraction (concentric and eccentric) will be controlled by an electronic metronome.
Maximal voluntary isometric contraction of knee extensors change after eight and sixteen weeks | Baseline, 8 week and 16 week
  The curve of maximum isometric muscle strength of knee extension will be collected at the same time as the eletromiography signal by dynamometer (MIOTEC, Porto Alegre, Brasil) connected to the electromyography. The subjects will receive instruction to exert maximal strength possible as fast as was possible when extending both knees. The subjects will have three attempts at obtaining the maximal voluntary contraction (MVC) of the knee extensors, each lasting 5 s.
Maximum muscular activity of vastus lateralis and rectus femoris change after eight and sixteen weeks | Baseline, 8 week and 16 week
  The maximal neuromuscular activity of agonist knee extensors muscles will be evaluate using surface electromyography (RMS values) on the vastus lateralis (VL) and rectus femoris (RF). Electrodes were positioned on the muscular belly in a bipolar configuration in parallel with the orientation of the muscle fibers, according to SENIAM project (www.seniam.org). To ensure the same electrode position in subsequent tests, the right thigh of each subject will be map out for the position of the electrode moles and small angiomas by marking on transparent paper.
Muscle thickness and echo intensity of knee extensors change after eight and sixteen weeks | Baseline, 8 week and 16 week
  Echo intensity and muscle thickness measures will be performed using ultrasound equipment (TOSHIBA-Tosbee/SSA-240A, Japan), with evaluation image in B-mode. Cross-sectional images will be obtained in the muscles of rights lower limbs: vastus lateralis, vastus medialis, vastus intermedius and rectus femoris. The images will be made in the vastus lateralis, vastus intermedius and rectus femoris (midway between the edge of the lateral condyle of the femur and the tip of the greater trochanter) and in the vastus medialis (20% between the edge of the lateral condyle of the femur and the tip of the greater trochanter). To ensure the same probe position in subsequent tests, the right thigh of each subject will be map out for the position of the transductor and small angiomas by marking on transparent paper.

SECONDARY OUTCOMES:
Dynamic muscular resistance change after sixteen weeks | Baseline and 16 week
  Dynamic muscular resistance will be evaluate during the bilateral knee extensors and free-weight barbell bilateral elbow flexors exercises using a load corresponding to 60% of the 1RM.
Cardiorespiratory Fitness evaluation change after sixteen weeks | Baseline and 16 week
  Protocol on the treadmill to determine the peak oxygen uptake change (VO2peak).
Cardiorespiratory Fitness evaluation change after sixteen weeks | Baseline and 16 week
  Protocol on the treadmill to determine the first ventilatory threshold.
Cardiorespiratory Fitness evaluation change after sixteen weeks | Baseline and 16 week
  Protocol on the treadmill to determine the second ventilatory threshold.
Heart rate change after sixteen weeks | Baseline and 16 week
  Heart rate resting.
Blood pressure change after sixteen weeks | Baseline and 16 week
  Resting blood pressure
Functional capacity change after sixteen weeks | Baseline and 16 week
  Tests: 30-Second Chair Stand.
Functional capacity change after sixteen weeks | Baseline and 16 week
  Test: 8-Foot Up-and-Go.
Functional capacity change after sixteen weeks | Baseline and 16 week
  Test: Chair sit-and-reach.
Functional capacity change after sixteen weeks | Baseline and 16 week
  Test: 6-Minute Walk
Functional capacity change after sixteen weeks | Baseline and 16 week
  Test: 8-Foot Up-and-Go during the dual-task condition
Quality of Life change after sixteen weeks (Score) | Baseline and 16 week
  World Health Organization Quality of Life - WHOQOL-bref. Scores range from 0 to 100 (0 being the lowest score possible). Higher values represent a better outcome.
Quality of Life change after sixteen weeks (Score) | Baseline and 16 week
  World Health Organization Quality of Life - WHOQOL-old. Scores can range from 24 to 120. Higher values represent better quality of life.
Cognitive function change after sixteen weeks (Score) | Baseline and 16 week
  Mini mental state examination The questionnaire consists of two parts, one that covers orientation, memory and attention (21 points). The second discusses specific skills such as naming and understanding (9 points). The scores range from 0 to 30. Higher values represent a better outcome.
Occurrence of low back pain change after sixteen weeks (%) | Baseline and 16 week
  Semi-structured questionnaire Percentage of occurrence of low back pain (higher values represent higher occurrence of low back pain).
Intensity of low back pain change after sixteen weeks (Scale) | Baseline and 16 week
  Semi-structured questionnaire. Numerical pain scale 0 (no pain) to 10 (worst pain possible).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Pinto, Phd, Principal Investigator — UFPel
Locations (1):
- Universidade Federal de Pelotas, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Hafele MS, Alberton CL, Hafele V, Schaun GZ, Nunes GN, Calonego C, Castro TF, Andrade LS, Pinto SS. Water-Based Training Programs Improve Functional Capacity, Cognitive and Hemodynamic Outcomes? The ACTIVE Randomized Clinical Trial. Res Q Exerc Sport. 2023 Mar;94(1):24-34. doi: 10.1080/02701367.2021.1935433. Epub 2022 Mar 16. PMID 35294330
- [Derived] Hafele MS, Alberton CL, Schaun GZ, Hafele V, Nunes GN, Andrade LS, Pinto SS. Quality of life responses after combined and aerobic water-based training programs in older women: a randomized clinical trial (ACTIVE Study). Aging Clin Exp Res. 2022 May;34(5):1123-1131. doi: 10.1007/s40520-021-02040-5. Epub 2022 Jan 13. PMID 35023049